CLINICAL TRIAL: NCT00001624
Title: Effect of Insulin on Endothelin-Dependent Vascular Tone in the Forearm Circulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970100; 97-H-0100
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-02

CONDITIONS: Hyperinsulinemia
Keywords: BQ-123; Endothelin; Insulin; Plethysmography; Vasoconstriction; Healthy Volunteer
MeSH Terms: conditions — Hyperinsulinism; Insulin Resistance | interventions — Insulin

INTERVENTIONS:
Drug: Insulin

SUMMARY:
Previous studies have shown that insulin may stimulate the release of endothelin (ET) from endothelial cells. This mechanism may contribute to the adverse vascular effects determined by chronic hyperinsulinemia. The aim of this study will be to evaluate the effect of local hyperinsulinemia on ET activity in the forearm circulation. To this purpose, we will assess the forearm blood flow response to ET receptor antagonism in control conditions and during intraarterial infusion of insulin. We will also measure changes in plasma ET-1 levels in response to the different pharmacological stimuli.

DETAILED DESCRIPTION:
Previous studies have shown that insulin may stimulate the release of endothelin (ET) from endothelial cells. This mechanism may contribute to the adverse vascular effects determined by chronic hyperinsulinemia. The aim of this study will be to evaluate the effect of local hyperinsulinemia on ET activity in the forearm circulation. To this purpose, we will assess the forearm blood flow response to ET receptor antagonism in control conditions and during intraarterial infusion of insulin. We will also measure changes in plasma ET-1 levels in response to the different pharmacological stimuli.

ELIGIBILITY:
Between 40-65 years old.

No medications.

No medical problems.

No serum cholesterol levels below 200 mg/dl.

No contraceptives.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16
Dates: Start 1997-03; Study Completion 2000-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Haynes WG, Webb DJ. Contribution of endogenous generation of endothelin-1 to basal vascular tone. Lancet. 1994 Sep 24;344(8926):852-4. doi: 10.1016/s0140-6736(94)92827-4. PMID 7916401
- [Background] Donckier J, Stoleru L, Hayashida W, Van Mechelen H, Selvais P, Galanti L, Clozel JP, Ketelslegers JM, Pouleur H. Role of endogenous endothelin-1 in experimental renal hypertension in dogs. Circulation. 1995 Jul 1;92(1):106-13. doi: 10.1161/01.cir.92.1.106. PMID 7788903